CLINICAL TRIAL: NCT00251654
Title: Complications and Adverse Effects in Continuous Peripheral Regional Anesthesia Results of Investigations on 3,491 Catheters
Brief Title: Complications and Adverse Effects in Continuous Peripheral Regional Anesthesia
Status: Completed | Type: Observational
Sponsor: Rechbergklinik Bretten (Other)
Collaborators: BG Unfallklinik Murnau (Other)
Responsible Party: Dr. M. Neuburger, OrtenauKlinikum Achern
Other Study IDs: MRA001
Record Dates: First submitted 2005-11-09; First posted 2005-11-10 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-09

CONDITIONS: Infection; Inflammation; Adverse Effects
Keywords: complications; adverse events; regional anesthesia; adverse effects
MeSH Terms: conditions — Infections; Inflammation | interventions — Anesthesia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: perineural block (anesthesia) — continuous peripheral regional anesthesia ropivacaine 0.33% for 3 to 5 days

SUMMARY:
The investigators prospectively document infectious, neurological, and other complications or adverse events occurring during peripheral regional anesthesia via a catheter using computer-based data recording.

DETAILED DESCRIPTION:
Perineural blocks with catheter placement are more and more frequently used. Few data dealing with infectious complications of perineural catheters exist. We assess incidence and localization of infectious complications of perineural catheters by means of computerized data acquisition. We prospectively evaluate perineural catheters placed at different sites for regional anesthesia and postoperative analgesia. The catheters were placed under standardized sterile conditions by using the nerve stimulator technique. Local inflammation is defined as the presence of at least two of the three signs: redness, pain on pressure or swelling. Infection is defined as the presence of at least two of the following criteria: pus at the catheter insertion site, fever, increased CRP and/or leukocytes requiring antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving perineural blocks via catheter

Exclusion criteria:

* None

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving perineural blocks via catheter ASA 1 to 4
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Actual)
Dates: Start 2002-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Büttner, MD, Study Chair — BG Unfallklinik Murnau
Locations (1):
- BG Unfallklinik, Murnau am Staffelsee, Bavaria, Germany

REFERENCES:
- [Result] Neuburger M, Breitbarth J, Reisig F, Lang D, Buttner J. [Complications and adverse events in continuous peripheral regional anesthesia Results of investigations on 3,491 catheters]. Anaesthesist. 2006 Jan;55(1):33-40. doi: 10.1007/s00101-005-0920-4. German. PMID 16193317
- [Result] Neuburger M, Buttner J, Blumenthal S, Breitbarth J, Borgeat A. Inflammation and infection complications of 2285 perineural catheters: a prospective study. Acta Anaesthesiol Scand. 2007 Jan;51(1):108-14. doi: 10.1111/j.1399-6576.2006.01173.x. Epub 2006 Nov 1. PMID 17073856
- [Result] Neuburger M, Reisig F, Zimmermann L, Buttner J. [Infection control in continuous peripheral regional anesthesia. Clinical study on disinfection time and subcutaneous tunneling in interscalene plexus anesthesia]. Anaesthesist. 2009 Aug;58(8):795-9. doi: 10.1007/s00101-009-1586-0. German. PMID 19669706